CLINICAL TRIAL: NCT04811287
Title: Utilizing Platelet-Rich Plasma as an Adjuvant to Carpal Tunnel Release for Severe Carpal Tunnel Syndrome
Brief Title: PRP as Adjuvant Treatment to CTR for Severe CTS Tunnel Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Fredericson, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Fredericson, MD, Professor of Orthopaedic Surgery, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59044
Record Dates: First submitted 2021-03-10; First posted 2021-03-23 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome; PRP
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using permuted block randomization predetermined by our dedicated orthopedic biostatistician into two study groups: those that undergo CTR with adjuvant intra-operative PRP and those that undergo CTR without adjuvant PRP.
Who Masked: Participant
Masking Description: See Model Description above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CTR with PRP (Active Comparator): Carpal tunnel release with adjuvant platelet-rich plasma.
  Interventions: Device: Carpal Tunnel Release with Platelet-Rich Plasma
- CTR without PRP (Placebo Comparator): Carpal tunnel release without adjuvant platelet-rich plasma.
  Interventions: Procedure: Carpal Tunnel Release without Platelet-Rich Plasma

INTERVENTIONS:
Device: Carpal Tunnel Release with Platelet-Rich Plasma — CTR is performed with adjuvant PRP placed intra-operatively.
  Arms: CTR with PRP
Procedure: Carpal Tunnel Release without Platelet-Rich Plasma — CTR is performed without adjuvant PRP placed intra-operatively.
  Arms: CTR without PRP

SUMMARY:
This study assesses the potential benefit of adjuvant platelet-rich plasma (PRP) with carpal tunnel release (CTR) for patients with severe carpal tunnel syndrome (CTS). CTR is a rather common procedure performed and seems to be quite effective for those with moderate CTS, but a number of patients with severe CTS do not have quite the same response post-CTR. The investigators will recruit patients who fall into the severe CTS category and compare CTR with and without adjuvant PRP to see if PRP can improve outcomes of this common surgery.

DETAILED DESCRIPTION:
1. Study team recruits patients with severe CTS who meet inclusion and exclusion criteria in an outpatient hand surgery clinic. Patients will be consented by the research team if the patient agrees to participate in the research study.
2. This will be a single blinded study, and participants will have an equal chance to be placed in either group. Participants will be randomized using permuted block randomization predetermined by our dedicated orthopedic biostatistician into two study groups: those that undergo CTR with adjuvant intra-operative PRP and those that undergo CTR without adjuvant PRP. All participants will have a pre-operative electromyography/nerve conduction study (EMG/NCS).
3. Primary outcome measures (BCTQ and grip strength), and secondary outcome measures (PROMIS; 2 point discrimination - thumb, index finger and middle finger; key pinch; 3 finger pinch; and EMG/NCS results) will be collected and stored in REDCap at initial visit. BCTQ and PROMIS will actually be available online for patient to complete at the patient's convenience.
4. Patients will undergo CTR with or without adjuvant PRP (based on assigned study group). Patients will not know which group the subject is in (single blinded).
5. BCTQ and PROMIS will be collected online at 3 months and 6 months post-operatively. EMG/NCS will only be performed preoperatively and at 6 months post-operatively in the Sports Medicine clinic. At the 6-month visit, the investigators will also collect data on 2 point discrimination, grip strength, key pinch, and 3 finger pinch.
6. The investigators will store data in REDCap.
7. Data will be analyzed with the assistance of our biostatistician, and results will be written up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 18 years and up.
2. Diagnosed with severe CTS based on EMG/NCS, meaning those with evidence of axonal loss (absent or low amplitude median sensory nerve action potential and/or absent or low amplitude median motor nerve action potential and/or evidence of abnormal spontaneous activity, reduced recruitment, or motor unit action potential changes on needle EMG of median innervated muscles).

Exclusion Criteria:

1. Younger than age 18 years (minor status).
2. Diagnosed with concomitant peripheral neuropathy.
3. Previous CTR on the affected side.
4. Have contraindications to PRP (platelet dysfunction syndrome, critical thrombocytopenia, hemodynamic instability, septicemia, local infection at site of procedure, consistent use of NSAIDs within 48 hours of procedure, steroid injection at treatment site within 1 month, systemic use of steroids within 2 weeks, tobacco use, recent fever or illness, or cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | up to 1 month pre-op
  Patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome.
Boston Carpal Tunnel Questionnaire | 3 months post-op
  Patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome.
Boston Carpal Tunnel Questionnaire | 6 months post-op
  Patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome.
Grip Strength | up to 1 month pre-op
  Measured with a dynamometer.
Grip Strength | 6 months post-op
  Measured with a dynamometer.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | up to 1 month pre-op
  Computer adaptive test developed to improve precision and reduce question burden for upper extremity conditions such as carpal tunnel syndrome.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 3 months post-op
  Computer adaptive test developed to improve precision and reduce question burden for upper extremity conditions such as carpal tunnel syndrome.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 6 months post-op
  Computer adaptive test developed to improve precision and reduce question burden for upper extremity conditions such as carpal tunnel syndrome.
2 Point Discrimination at Thumb | up to 1 month pre-op
  Minimal distance that the patient feels 2 separate points of touch.
2 Point Discrimination at Thumb | 6 months post-op
  Minimal distance that the patient feels 2 separate points of touch.
2 Point Discrimination at Index Finger | up to 1 month pre-op
  Minimal distance that the patient still feels 2 separate points of touch.
2 Point Discrimination at Index Finger | 6 months post-op
  Minimal distance that the patient still feels 2 separate points of touch.
2 Point Discrimination at Middle Finger | up to 1 month pre-op
  Minimal distance that the patient still feels 2 separate points of touch.
2 Point Discrimination at Middle Finger | 6 months post-op
  Minimal distance that the patient still feels 2 separate points of touch.
Key Pinch | up to 1 month pre-op
  Measured with a pinch meter.
Key Pinch | 6 months post-op
  Measured with a pinch meter.
3 Finger Pinch | up to 1 month pre-op
  Measured with a pinch meter.
3 Finger Pinch | 6 months post-op
  Measured with a pinch meter.
Median Motor Latency | up to 1 month pre-op
  From EMG/NCS data.
Median Motor Latency | 6 months post-op
  From EMG/NCS data.
Median Motor Amplitude | up to 1 month pre-op
  From EMG/NCS data.
Median Motor Amplitude | 6 months post-op
  From EMG/NCS data.
Median Sensory Latency | up to 1 month pre-op
  From EMG/NCS data.
Median Sensory Latency | 6 months post-op
  From EMG/NCS data.
Median Sensory Amplitude | up to 1 month pre-op
  From EMG/NCS data.
Median Sensory Amplitude | 6 months post-op
  From EMG/NCS data.
EMG of Abductor Pollicis Brevis | up to 1 month pre-op
  From EMG/NCS data - looking at spontaneous activity.
EMG of Abductor Pollicis Brevis | 6 months post-op
  From EMG/NCS data - looking at spontaneous activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trull-Ahuir C, Sala D, Chismol-Abad J, Vila-Caballer M, Lison JF. Efficacy of platelet-rich plasma as an adjuvant to surgical carpal ligament release: a prospective, randomized controlled clinical trial. Sci Rep. 2020 Feb 7;10(1):2085. doi: 10.1038/s41598-020-59113-0. PMID 32034241